CLINICAL TRIAL: NCT00071877
Title: A Clinical Trial of Replagal Enzyme Replacement Therapy in Children Ages 7 - 17 Years With Fabry Disease
Brief Title: An Open-Label Clinical Trial of Replagal Enzyme Therapy in Children Ages 7-17 Years With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040029; 04-N-0029
Record Dates: First submitted 2003-11-03; First posted 2003-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-06

CONDITIONS: Fabry Disease
Keywords: Lysosomal Disease; Hypohidrosis; Pain; Neuropathy; X-Linked; Fabry Disease; Children
MeSH Terms: conditions — Fabry Disease; Hypohidrosis; Pain | interventions — agalsidase alfa

INTERVENTIONS:
Drug: Replagal

SUMMARY:
This study will evaluate the safety of multiple biweekly intravenous doses of Replagal over 26 weeks in 25 children with Fabry disease and the way in which that agent can improve the health of this patient population. Fabry disease is a genetic disorder inherited as an X-linked recessive trait. It causes a deficiency in the enzyme alpha galactosidase, which normally breaks down a lipid, or fatty substance, called ceramidetrihexosidase, a building block in all cells of the body.

The deficiency in breaking down the lipid eventually causes that lipid to accumulate and injure cells. Problems in the blood vessels, kidneys, heart, and nerves are the result. The disease typically occurs in childhood or adolescence, with repeated episodes of severe pain in the extremities and other symptoms. There is no definitive treatment, but pain management is important in caring for patients with Fabry disease. Although it is not known exactly how lipid accumulation brings about such problems, studies of another lipid storage disorder, Gaucher's disease, have shown that the illness can be reversed if the lipid is removed when an appropriate enzyme, Replagal, is given intravenously. In this study, the gene response of the body's cells to Fabry disease will be described, as will any gene responses that change when the enzyme is used.

Patients 7 to 17 years of age who have Fabry disease may be eligible for this study. They will undergo the following tests and procedures:

* Physical examination.
* Neurological examination.
* Vital signs.
* Urinalysis.
* Blood tests to determine complete blood count and chemistries.
* Questionnaire on pain.
* Tests pertaining to sweating.
* Electrocardiogram.
* Doppler blood flow study.
* Diary for recording symptoms and the use of pain medications.

Participants will go through the evaluation, over a period of about 5 days, either as an inpatient or outpatient. Participants will receive an intravenous infusion of Replagal every other week, at the dose of 0.2 mg/kg of body weight. Vital signs will be measured before the infusion and immediately and after and 1 hour afterward. There will be careful monitoring for allergic reactions and side effects. The infusion time takes approximately 40 minutes.

This study will last 6 months, with the possibility of being extended another 6 months-a maintenance study in which patients will continue to receive Replagal at the same dose every 2 weeks.

DETAILED DESCRIPTION:
The objectives of this clinical trial are to evaluate: 1) the safety of multiple biweekly (i.e. every other week) intravenous (IV) doses of Replagal over 26 weeks in 25 children ages 7-17 years old with Fabry Disease, and 2) the pharmacokinetics of Replagal in this patient population. Safety will be determined by standard clinical and laboratory measurements.

ELIGIBILITY:
INCLUSION CRITERIA:

Male hemizygote with Fabry Disease as documented by clinical evidence and by laboratory evidence of alpha-galactosidase A deficiency.

Or

Female heterozygote with Fabry Disease as documented by gene analysis showing a mutation of the alpha-galactosidase A gene. Female patients of child-bearing potential must have a negative pregnancy test at baseline and agree to the use of effective contraception such as oral contraceptive or double barrier method for study entry and while participating in the study.

7-17 years of age.

Adequate general health (as determined by the investigators) to undergo the specified phlebotomy regimen and protocol related procedures.

The child must assent to participate in the protocol and the parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee (IRB/IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed with the child and the child's parent(s) or legal guardian(s).

EXCLUSION CRITERIA:

Patient has previously participated in a multi-dose clinical study of an investigational therapeutic agent for Fabry Disease.

Patient and/or the patient's parent(s) or legal guardian(s) are unable to understand the nature, scope, and possible consequences of the study.

Patient is unable to comply with the protocol, e.g., uncooperative with protocol schedule, refusal to agree to all of the study procedures, inability to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the investigator or the medical monitor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2003-10; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Brady RO, Gal AE, Bradley RM, Martensson E, Warshaw AL, Laster L. Enzymatic defect in Fabry's disease. Ceramidetrihexosidase deficiency. N Engl J Med. 1967 May 25;276(21):1163-7. doi: 10.1056/NEJM196705252762101. No abstract available. PMID 6023233
- [Background] Kahn P. Anderson-Fabry disease: a histopathological study of three cases with observations on the mechanism of production of pain. J Neurol Neurosurg Psychiatry. 1973 Dec;36(6):1053-62. doi: 10.1136/jnnp.36.6.1053. PMID 4204059
- [Background] Kaye EM, Kolodny EH, Logigian EL, Ullman MD. Nervous system involvement in Fabry's disease: clinicopathological and biochemical correlation. Ann Neurol. 1988 May;23(5):505-9. doi: 10.1002/ana.410230513. PMID 3133979